CLINICAL TRIAL: NCT02644525
Title: A Double-blinded, Randomized, Placebo-Controlled Dose Escalation Study to Examine the Efficacy and Microfilaricidal Kinetics and Safety of Imatinib for the Treatment of Loa Loa (A Pilot Study)
Brief Title: Efficacy and Microfilaricidal Kinetics of Imatinib for the Treatment of Loa Loa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Planned interim analysis demonstrated futility of intervention
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999916042; 16-I-N042
Record Dates: First submitted 2015-12-31; First posted 2016-01-01 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2021-03

CONDITIONS: Loiasis
Keywords: Cameroon; Filaricidal; Randomized; Blinded; Diethylcarbamazine; Imatinib; Loa loa
MeSH Terms: conditions — Loiasis | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects given vitamin placebo
  Interventions: Drug: Placebo
- Imatinib 200mg (Experimental): Subjects given a single dose of imatinib 200mg PO
  Interventions: Drug: Imatinib Mesylate
- Imatinib 400mg (Experimental): Subjects given a single dose of imatinib 400mg PO
  Interventions: Drug: Imatinib Mesylate
- Imatinib 600mg (Experimental): Subjects given a single dose of imatinib 600mg PO
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — A single dose of imatinib 200mg PO is given
  Other Names: Gleevec
  Arms: Imatinib 200mg
Drug: Imatinib Mesylate — A single dose of imatinib 400mg PO is given
  Other Names: Gleevec
  Arms: Imatinib 400mg
Drug: Imatinib Mesylate — A single dose of imatinib 600mg PO is given
  Other Names: Gleevec
  Arms: Imatinib 600mg
Drug: Placebo — A single dose of placebo pill is given
  Arms: Placebo

SUMMARY:
Background:

Many people who live in west or central Africa are at risk for infection from a very small worm called Loa loa. This infection is acquired through the bite of a fly. Baby worms called microfilariae live in the blood. The infection most commonly causes skin itching, mild temporary limb swelling, and sometimes a adult worm can be seen in the white of the eye of an infected individual. Very rarely, people with this infection can develop problems with the kidneys and heart as a result of the worm's effect on the immune system. Because the vast majority of people with the infection have minimal symptoms, people in Cameroon usually do not get treated. But infection with Loa loa can cause serious problems in people who are being treated for infections with other parasites (namely, river blindness and lymphatic filariasis). Researchers want to find out of a drug called imatinib can treat Loa loa infection so that patients with this infection can safely receive other drugs to cure river blindness and lymphatic filariasis. Researchers believe imatinib can be a safe drug to use on Loa loa, because in the lab this drug kills the worms slowly, whereas other drugs which can cause treatment reactions usually kill the worms very quickly.

Objective:

To test if imatinib can treat Loa loa infection by killing the worms slowly.

Eligibility:

People ages 18-65 with non-severe Loa loa infection who are otherwise healthy

Design:

Participants will be screened with a physical exam and blood and urine tests.

Participants will have a baseline visit. This will include a physical exam and blood and urine tests. It may include a stool sample. Participants will be randomly assigned to get 1 dose of either imatinib or a placebo.

Participants will return to the clinic every day for 1 week, then once a week for 3 weeks. Visits will include a physical exam and blood tests. They will have urine tests in the first week.

Participants will have follow-up visits 3, 6, and 12 months after taking the imatinib or placebo. These include a physical exam and blood tests. They may include urine and stool samples.

If participants develop side effects, they will be treated for them.

DETAILED DESCRIPTION:
With the discovery that people experiencing severe treatment reactions following mass drug administration (MDA) with ivermectin for onchocerciasis and lymphatic filariasis control were co-infected with Loa loa, there has been a need for new filaricidal drugs. Currently, Loa loa infection, considered relatively nonpathogenic, is not treated in endemic areas. However, because treatment for Loa loa can result in toxicity in people who are being concurrently treated for onchocerciasis and lymphatic filariasis, finding a new treatment for Loa loa has become a priority. Imatinib has recently been shown to be microfilaricidal in vitro at concentrations physiologically achievable after a single oral dose in humans. The current standard in loiasis treatment outside of endemic areas is to treat those with low microfilarial (MF) levels (less than approximately 8,000MF/mL) with diethylcarbamazine (DEC). However, at high MF concentrations (>20,000 MF/mL) serious side effects including encephalopathy and death have occurred with administration of DEC or ivermectin, a widely distributed microfilaricide throughout Africa. In endemic areas, this risk is avoided by not treating loiasis altogether. The adverse reactions are believed to be due release of a large antigen load due to rapid killing of large numbers of MF. The rapidity of killing is believed to be the main driver of these reactions seen at high MF counts. The purpose of this study is to assess how imatinib acts as a slow microfilaricide at levels (<2,500 MF/mL) that have been safely treated previously with DEC and ivermectin. We aim to perform a dose escalation study to identify the minimum single oral dose that will be effective as a slow microfiaricidal drug against Loa loa. If imatinib is found to be effective and have kinetics which favor slow microfilarial killing, then this can serve as the basis for a larger study in which patients with very high microfilarial loads would be treated, as this is the at risk population in current MDA campaigns. This is a double blind, randomized, pilot phase 2 dose-escalation trial. Subjects will receive a dose of imatinib at 200, 400 or 600 (n = 5 each). Symptoms and blood microfilarial concentration will be assessed at baseline, daily for the first 7 days, then weekly for the next 21 days, then at 3, 6, and 12 months. These will be compared against an untreated placebo-controlled group of 5 subjects who will have the same data collected at these respective days.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years old and less than or equal to 65 years
  2. Loa loa microfilaremia >500 MF/mL and <2500 MF/mL at screening visit.
  3. Subject has the capacity to understand the potential risks and benefits and consents to protocol indicated blood draws and follow up visits.

EXCLUSION CRITERIA:

1. Women under 45 years of age, or over 45 years of age with a menstrual period in the preceding 12 months.
2. Currently breastfeeding
3. Currently taking daily medications
4. Known chronic medical conditions, including but not limited to diabetes, renal failure, liver disease, seizure disorder, HIV, malignancy, psychiatric disorder, or any conditions which within the investigators judgement are deemed to be clinically significant.
5. W. bancrofti serologic positivity against Wb123
6. O. volvulus serologic positivity against Ov16
7. HIV by history or clinical signs of HIV/AIDS (e.g. oral thrush, oral/skin lesions of Kaposi s sarcoma, etc.)
8. Any of the following lab abnormalities: Creatinine >1.5, Platelets <100,000/mL, Hemoglobin <12g/dL, alanine aminotransferase or aspartate aminotransferase >60 U/L, total bilirubin >1.7mg/dL, absolute neutrophil count equal to or less than 1500/mm(3).
9. Any condition that, in the opinion of the PI, may substantially increase the risk of participation, including any contraindication to imatinib.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise M O'Connell, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Centre de Recherche sur les Filarioses et Autres Maladies Tropicales, Mbalmayo, Cameroon

REFERENCES:
- [Background] Boussinesq M, Gardon J, Gardon-Wendel N, Chippaux JP. Clinical picture, epidemiology and outcome of Loa-associated serious adverse events related to mass ivermectin treatment of onchocerciasis in Cameroon. Filaria J. 2003 Oct 24;2 Suppl 1(Suppl 1):S4. doi: 10.1186/1475-2883-2-S1-S4. PMID 14975061
- [Background] O'Connell EM, Nutman TB. Reduction of Loa loa Microfilaremia with Imatinib - A Case Report. N Engl J Med. 2017 Nov 23;377(21):2095-2096. doi: 10.1056/NEJMc1712990. No abstract available. PMID 29166233
- [Background] Twum-Danso NA. Loa loa encephalopathy temporally related to ivermectin administration reported from onchocerciasis mass treatment programs from 1989 to 2001: implications for the future. Filaria J. 2003 Oct 24;2 Suppl 1(Suppl 1):S7. doi: 10.1186/1475-2883-2-S1-S7. PMID 14975064

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 5 subjects given placebo as a single dose
- Imatinib 200mg: Participants given a single dose of 200mg PO imatinib
- Imatinib 400mg: Participants given a single dose of 400mg PO imatinib
- Imatinib 600mg: Participants given a single dose of 600mg PO imatinib
Period: Group 1
Arm/Group | Placebo | Imatinib 200mg | Imatinib 400mg | Imatinib 600mg
Started | 2 | 5 | 0 | 0
Completed | 2 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Group 2
Arm/Group | Placebo | Imatinib 200mg | Imatinib 400mg | Imatinib 600mg
Started | 2 | 0 | 5 | 0
Completed | 2 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Group 3
Arm/Group | Placebo | Imatinib 200mg | Imatinib 400mg | Imatinib 600mg
Started | 1 | 0 | 0 | 5
Completed | 1 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Imatinib 200mg: 5 subjects given 200mg PO imatinib as a single dose
- Imatinib 400mg: 5 subjects given 400mg PO imatinib as a single dose
- Imatinib 600mg: 5 subjects given 600mg PO imatinib as a single dose
- Total: Total of all reporting groups
Arm/Group | Placebo | Imatinib 200mg | Imatinib 400mg | Imatinib 600mg | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [41 to 64] | 51 [32 to 64] | 50 [19 to 65] | 45 [29 to 65] | 49 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 2 | 3
  Male | 4 | 5 | 5 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 5 | 5 | 20
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Cameroon | 5 | 5 | 5 | 5 | 20
Loa loa mid-day blood microfilariae count [Geometric Mean (Full Range); unit: microfilariae/mL] | 1447 [520 to 3120] | 1329 [760 to 2340] | 2154 [1000 to 6540] | 1328 [640 to 3060] | 1532 [520 to 6540]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Baseline Loa Loa Microfilariae
Description: Percent of baseline Loa loa microfilariae as determined by concentrated peripheral blood smear. Daily measurements will be taken the first week, followed by measurements at day 14 and day 21
Time Frame: Days 1-7, 14, 21
Population: In a two cases (Day 2 for Imatinib 200mg, Day 7 for Imatinib 400mg), some values were missing.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline microfilariae
Groups:
- Placebo: Single dose of placebo
- Imatinib 200mg: Single dose of imatinib 200mg po
- Imatinib 400mg: Single dose of imatinib 400mg po
- Imatinib 600mg: Single dose of imatinib 600mg po
Arm/Group | Placebo | Imatinib 200mg | Imatinib 400mg | Imatinib 600mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
percentage of baseline microfilariae
  Day 1 | 88.7 [52.2 to 150.8] | 114.5 [81.2 to 161.4] | 104.7 [82.4 to 133.1] | 102.2 [56.0 to 186.5]
  Day 2: number analyzed (Participants) | 5 | 4 | 5 | 5
  Day 2 | 88.1 [61.7 to 125.7] | 96.8 [48.0 to 195.5] | 98.0 [70.6 to 135.9] | 97.8 [53.3 to 179.5]
  Day 3 | 84.6 [49.6 to 144.4] | 102.8 [70.8 to 149.1] | 84.0 [51.9 to 136.0] | 84.8 [61.4 to 117.0]
  Day 4 | 73.3 [46.5 to 115.5] | 108.5 [72.3 to 163.0] | 59.7 [23.5 to 151.7] | 88.1 [62.1 to 125.1]
  Day 5 | 79.9 [40.6 to 157.2] | 95.5 [67.5 to 135.2] | 76.9 [22.7 to 260.5] | 89.1 [55.8 to 142.3]
  Day 6 | 80.4 [50.3 to 128.5] | 107.0 [72.4 to 158.0] | 62.3 [16.8 to 230.8] | 84.1 [49.1 to 144.1]
  Day 7: number analyzed (Participants) | 5 | 5 | 1 | 5
  Day 7 | 76.9 [52.2 to 113.2] | 78.9 [41.9 to 148.5] | 136.0 [NA to NA] — missing data, not enough non-missing data to calculate confidence interval | 83.3 [70.2 to 98.9]
  Day 14 | 100.6 [52.2 to 193.7] | 83.7 [51.9 to 135.0] | 81.8 [30.8 to 217.4] | 94.4 [65.2 to 136.6]
  Day 21 | 66.8 [38.1 to 116.9] | 86.5 [36.8 to 203.2] | 107.6 [66.1 to 175.2] | 97.4 [73.5 to 129.1]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Common Terminology Criteria for Adverse Events v5.0. Refer to protocol for schedule of labs and history and physical exams to collect this data over 3 months.
Arm/Group | Placebo | Imatinib 200mg | Imatinib 400mg | Imatinib 600mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 2/5 | 1/5
Other Adverse Events (participants affected / at risk) | 4/5 | 5/5 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Imatinib 200mg (N=5) | Imatinib 400mg (N=5) | Imatinib 600mg (N=5)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3 Systolic Blood Pressure Hypertension
Neutropenia (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Grade 3 neutropenia
Pulmonary embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Imatinib 200mg (N=5) | Imatinib 400mg (N=5) | Imatinib 600mg (N=5)
Headache (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 2 (2) | 3 (4)
Anorexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1)
Blood bilirubin increased (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (4) | 3 (5) | 3 (6) | 1 (2)
Hyponatremia (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Insomnia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphedema (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mild wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (5) | 4 (6) | 3 (4) | 3 (5)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 2 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (2)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT02644525/Prot_SAP_000.pdf
  • Informed Consent Form: English (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02644525/ICF_001.pdf